CLINICAL TRIAL: NCT06118866
Title: A Randomized, Multicenter, Double-blind, Placebo-Controlled Phase 2 Study to Evaluate the Safety, Tolerability and Efficacy in Male Androgenetic Alopecia Treated With HMI-115 Over a 24-Week Treatment Period
Brief Title: A Study to Assess the Efficacy and Safety of HMI-115 in Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Medicine (Nanjing) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMI-115AG201
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- placebo-Q2W (Placebo Comparator): placebo, 0mg/vials
  Interventions: Drug: placebo-Q2W
- HMI-115-120mg-Q4W (Active Comparator): HMI-115, 60mg/vials
  Interventions: Drug: HMI-115-120mg-Q4W
- HMI-115-240mg-Q4W (Active Comparator): HMI-115, 60mg/vials
  Interventions: Drug: HMI-115-240mg-Q4W
- HMI-115-240mg-Q2W (Active Comparator): HMI-115, 60mg/vials
  Interventions: Drug: HMI-115, 240mg-Q2W

INTERVENTIONS:
Drug: placebo-Q2W — placebo, 0mg，SC，Q2W，12 cycles
  Arms: placebo-Q2W
Drug: HMI-115-120mg-Q4W — HMI-115, 120mg，SC，Q4W，6 cycles(Placebo given in the second week of each cycle)
  Arms: HMI-115-120mg-Q4W
Drug: HMI-115-240mg-Q4W — HMI-115, 240mg，SC，Q4W，6 cycles(Placebo given in the second week of each cycle)
  Arms: HMI-115-240mg-Q4W
Drug: HMI-115, 240mg-Q2W — HMI-115, 240mg，SC，Q2W，12 cycles
  Arms: HMI-115-240mg-Q2W

SUMMARY:
To investigate the efficacy of HMI-115 compared to placebo in treating Androgenic Alopecia patients for 24 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Male subjects, between 18 and 65 years of age, inclusive, at the time of signing informed consent.
3. Clinical diagnosis of androgenetic alopecia. Male subjects who meet Norwood-Hamilton scales III vertex, IV and V .
4. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions, including having a small circle about 1 cm2 of hair clipped to approximate 1 mm in length and micro-dot-tattoo on the scalp of target area.
5. Subjects who are willing to keep the same hair color, refrain from hair weaving, and hair growth therapy and supplement (except for protocol specified IMP) during the study.
6. Subjects agree to use required birth control methods from signing the consent until 3 months after the last dose of IMP or complete whole study period whichever is longer.

Exclusion Criteria:

1. Subject with history of scalp radiation or surgery which could interfere study assessment (e.g., hair transplantation surgery).
2. Subject with history of scalp laser treatment within 6 months prior screening, including but not limited to, low level laser, and fractional laser, etc.
3. Subject with history of hair weaves within 3 months prior screening.
4. Subject has a current history of hyperthyroidism or uncontrolled hypothyroidism.
5. Subject has, in the Investigator's opinion, uncontrolled hypertension (systolic blood pressure [SBP] > 159 mmHg, diastolic blood pressure [DBP] > 99 mmHg).
6. Subject has any of the following conditions within 6 weeks prior to Screening:

   1. Myocardial infarction, stroke, unstable angina, or transient ischemic attack.
   2. Heart failure with classified as being in New York Heart Association Class III or IV.
7. Subject has high fever, major surgery, or ten percent or more weight decrease within three months before screening.
8. Subject with history of active malignancy (with or without systemic chemotherapy), except treated basal cell carcinoma of the skin (besides scalp).
9. Subject plans to schedule elective surgery during the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
The Rate of Target Arean Hair Count (TAHC) | 24 Weeks
  The mean change in TAHC of non-vellus from baseline

SECONDARY OUTCOMES:
Hair Growth State Assessed by Hair Growth Questionnaire Assessment (HGQA) | 6 weeks, 12 weeks, 18 weeks, 24 weeks, and 36 weeks
  To assess the hair growth by 7-question questionnaire and summary the number and percentage of subjects in each category for each HGQA question.
Target Area Hair Count (TAHC) change from baseline | 6 weeks, 12 weeks, 18 weeks, 24 weeks, and 36 weeks
  The mean change in TAHC of non-vellus from Baseline
Rate of Target Area Hair Width (TAHW) | 6 weeks, 12 weeks, 18 weeks, 24 weeks, and 36 weeks
  The mean change in TAHW of non-vellus from baseline
Investigator Global Assessment (IGA) | 6 weeks, 12 weeks, 18 weeks, 24 weeks, and 36 weeks
  Summary of subject number and percentage in each IGA category
Subject Self-Assessment (SSA) | 6 weeks, 12 weeks, 18 weeks, 24 weeks, and 36 weeks
  Summary of subject number and percentage in each SSA category
Norwood-Hamilton Grade change from baseline | 12 weeks, 24 weeks, and 36 weeks
  Summary of subject number and percentage in each grade of Norwood-Hamilton Scale
Frequencies and percentages of Adverse event (AE) | 36Weeks
  Frequency and percentages of subjects with treatment-emergent AE (TEAE) will be calculated and TEAE will be summarized by systematic organ classification (SOC), preferred term (PT), relationship to study treatment, maximum severity, whether resulting in death, whether resulting in study treatment discontinuation, belong to serious AE (SAE) or not, belong to events of special interest (AESI) or not.
Blood Pressure change from baseline | 36 Weeks
  Descriptive statistics summarizing changes in blood pressure (systolic and diastolic) will be compared between baseline levels and each predetermined time point.
Pulse change from baseline | 36 Weeks
  Descriptive statistics summarizing changes in pulse will be compared between baseline levels and each predetermined time point.
Body temperature change from baseline | 36 Weeks
  Descriptive statistics summarizing changes in body temperature will be compared between baseline levels and each predetermined time point.
Respiratory rate | 36 Weeks
  Descriptive statistics summarizing changes in respiratory rate will be compared between baseline levels and each predetermined time point.
Complete or brief physical examination, at a minimum of General appearance, HEENT (head, eyes, ears, nose, throat), Neck, Lung/pulmonary, Chest, Neurological or not, Extremities,ect.to assess the physical health state. | 36 Weeks
  Physical examination findings by body system will be summarized, presented with frequency counts and percentages. A complete or brief physical examination will be performed at Visit 1, Visit 2, End of Treatment Visit and Follow-up Visit. Height (cm) and weight (kg) will be measured and body mass index will be calculated and recorded at specified period.
Concomitant Medication | 36 Weeks
  Concomitant medication usage will be summarized by the number and proportion of subjects and classified by the World Health Organization Drug Dictionary (WHO DD) based on Anatomical Therapeutic Chemical Classification System (ATC) code level 3.
Change in twelve-lead electrocardiogram parameters | 36 Weeks
  Change in electrocardiogram parameters including heart rate (HR), QRS, RR, PR, and QT interval (QTcF and QTcB) relative to baseline will be summarized descriptively by visits and groups. The within-group changes from baseline to each visit will be summarized and will be compared with a paired t-test for continuous measurements. Subject number and percentage with other clinically significant electrocardiogram findings in each visit will be summarized by groups. A general assessment of the 12-lead electrocardiogram will be presented as normal, abnormal clinical significance, or abnormal no clinical significance.
Clinical laboratory tests of hematology | 36 Weeks
  Descriptive statistics summarizing changes in results of clinical laboratory tests of hematology from baseline levels at each predetermined time point. Shift tables for changes from baseline according to the normal minimum and maximum will be provided.
Clinical laboratory tests of coagulation | 36 Weeks
  Descriptive statistics summarizing changes in results of clinical laboratory tests of coagulation from baseline levels at each predetermined time point. Shift tables for changes from baseline according to the normal minimum and maximum will be provided.
Clinical laboratory tests of clinical chemistry | 36 Weeks
  Descriptive statistics summarizing changes in results of clinical laboratory tests of clinical chemistry from baseline levels at each predetermined time point. Shift tables for changes from baseline according to the normal minimum and maximum will be provided.
Clinical laboratory tests of urinalysis | 36 Weeks
  Descriptive statistics summarizing changes in results of clinical laboratory tests of urinalysis from baseline levels at each predetermined time point. Shift tables for changes from baseline according to the normal minimum and maximum will be provided.
Clinical laboratory tests of hormones | 36 Weeks
  Descriptive statistics summarizing changes in results of clinical laboratory tests of hormones from baseline levels at each predetermined time point. Shift tables for changes from baseline according to the normal minimum and maximum will be provided.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No